CLINICAL TRIAL: NCT01792011
Title: Accuracy and Utility of the Pleth Variability Index as a Predictor of Fluid Responsiveness During the Dissection and Anhepatic Phase of Liver Transplantation
Brief Title: Accuracy of the Pleth Variability Index to Predict Fluid Responsiveness in Liver Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Gulay ERDOGAN KAYHAN, MD,Asistant Professor Dr, Inonu University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: Institute of LLT
Record Dates: First submitted 2013-02-08; First posted 2013-02-15 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Hemodynamic Instability
Keywords: Elective living donor liver transplantation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PVI (Experimental): A new non-invasive device (Radical-7 pulse oximeter monitor, Masimo Corp.) has been introduced that continuously detects changes in the plethysmograph waveform and computes a Plethysmography Variability Index (PVI) reflecting alteration in preload and fluid management.
  Interventions: Device: PVI-guided fluid management

INTERVENTIONS:
Device: PVI-guided fluid management — In this study of 25 adult patients undergoing OLT, we prospectively record PVIwithin 5 minutes during dissection and anhepatic phase of OLT by Masimo pulse oximeter.In this study of 25 adult patients undergoing OLT, we prospectively record study data within 5 minutes during dissection and anhepatic phase of OLT. Study data included measurements of PVI,thermodilution cardiac output, Stroke volume variation (SVV) and Pulse pressure variation (PPV).

SUMMARY:
The aim of this study is to compare the accuracy of PVI (pleth variability index)

DETAILED DESCRIPTION:
The aim of this study is to compare the accuracy of PVI (pleth variability index)with other hemodynamic variability that measured with PİCCO (SVV, PPV, CVP,CI)to predict the response of cardiac index to volume replacement in patients undergoing liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Elective living donor liver transplantation,
* >18 years patients

Exclusion Criteria:

Patients with:

* Arrhythmia
* Reduced left ventricular function (EF<40%)
* Hepatocellular carcinoma
* Pulmonary hypertension
* Fulminant liver failure
* valvular heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
To test the ability of PVI to detect changes in preload during orthotopic liver transplantation | During dissection and anhepatic phase (3 months)
  PVI is a measure of the dynamic changes in perfusion index that occur during a complete respiratory cycle

CONTACTS AND LOCATIONS:
Overall Officials: Gulay Erdogan Kayhan, Dr, Study Chair — Inonu University Faculty of Medicine Anesthesiology and Reanimation Department
Locations (1):
- Inonu University Faculty of Medicine Department of Anesthesiology and Reanimation, Malatya, Turkey (Türkiye)